CLINICAL TRIAL: NCT00534300
Title: Intravenous Infusion of n-3 Polyunsaturated Fatty Acids and Ventricular Tachycardia in Patients With Implantable Cardioverter Defibrillator (ICD)
Brief Title: Intravenous n-3 Fatty Acids and Ventricular Tachycardia in Patients With Implantable Cardioverter Defibrillator (ICD)-Pacemaker
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Trine Madsen, Aalborg Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: IVN3ICD; EudraCT number: 2005-002386-37
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Ventricular Tachycardia; Sudden Cardiac Death
Keywords: ICD-pacemaker
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac | interventions — fish oil triglycerides; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Omegaven
- B (Placebo Comparator)
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Omegaven — Lipid emulsion (omegaven) for intravenous use, 100 ml (25 mL/h)
  Arms: A
Drug: Isotonic saline — Intravenous infusion, 100 mL, 25mL/h
  Arms: B

SUMMARY:
The long-chain n-3 polyunsaturated fatty acids (PUFA), eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), appear to offer protection against sudden cardiac death and ventricular arrhythmias. EPA and DHA are essential fatty acids which are incorporated into cellular membranes after regular ingestion of fatty fish or fish oil.

This study investigates a possible acute effect of intravenous infusion of n-3 PUFA on inducibility of ventricular tachycardia (VT) in patients with an ICD-pacemaker.

The hypothesis is that an acute rise in the concentration of n-3 PUFA in plasma will increase the electric stability of the myocardial cells, so that VT is more difficult to induce.

In a randomized, placebo-controlled, double-blind, crossover study, a lipid emulsion with a high content of n-3 PUFA (or placebo: isotonic saline) will be administered intravenously before a non-invasive electrophysiologic examination performed via the ICD and following a predefined protocol.

The main outcome is inducibility of VT. If sustained VT is induced in a patient after both n-3 PUFA and placebo, the strength of the required stimulus after n-3 PUFA and after placebo is compared.

ELIGIBILITY:
Inclusion Criteria:

* Sustained ventricular tachycardia (VT) inducible during primary electrophysiological study (before ICD implantation) and one of the following

  * Latest VT episode terminated by anti-tachycardia pacing (ATP)
  * VT induced during primary electrophysiological study terminated by ATP

Exclusion Criteria:

* Premenopausal women
* Allergy to fish or egg protein
* Blood pressure > 160/90 (treated or untreated)
* MI, PCI or CABG within the previous 6 months
* HbA1c > 10%
* ALT > 150 U/L
* INR > 3.5
* Plasma-potassium < 3.5 mmol/L
* Fasting triglycerides > 3 mmol/L
* Other serious illness
* Inability to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Inducibility of ventricular tachycardia | Hours

SECONDARY OUTCOMES:
Heart rate variability | Hours
Ventricular repolarization parameters | Hours
Concentration of n-3 fatty acids in plasma and platelet membranes | Hours

CONTACTS AND LOCATIONS:
Overall Officials: Trine Madsen, MD, Principal Investigator — Aalborg Hospital, Aarhus University Hospital, Denmark
Locations (1):
- Department of Cardiology, Aalborg Hospital, Aalborg, Denmark